CLINICAL TRIAL: NCT06288217
Title: Feasibility of Trigeminal and Vagus Nerve Stimulation in Subjects With Chronic Upper Extremity Deficits After Stroke
Brief Title: Non-invasive Trigeminal and Vagus Nerve Stimulation for Stroke Subjects With Chronic Upper Extremity Deficits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeuraStasis, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NS-CIP-001
Record Dates: First submitted 2024-02-17; First posted 2024-03-01 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stroke, Ischemic; Upper Extremity Paresis
MeSH Terms: conditions — Ischemic Stroke; Paresis | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Paired nTVNS Stimulation (Experimental): Non-invasive electrical stimulation of the trigeminal and vagus nerves will be delivered by the NeuraStasis Stimulator System. The non-invasive Stimulation Electrode is positioned on the head (forehead and in the ear). The operator controls the stimulation delivery through the accompanying Controller.
  Rehabilitation sessions begin with a stimulation tolerability assessment where the dose of therapy is selected. A 15-minute priming stimulation is delivered next, followed by the standard of care rehabilitation over the remaining session. During this rehabilitation paired nTVNS is delivered with repetitive motions.
  Interventions: Device: NeuraStasis Stimulator System (Non-Invasive Trigeminal and Vagus Nerve Stimulation); Other: Upper Limb Rehabilitation
- Sham Stimulation (Sham Comparator): For the active shame comparator group, the non-invasive Stimulation Electrode is positioned on the head (forehead and in the ear) as in the experimental group. The operator controls the stimulation delivery through the accompanying Controller.
  Rehabilitation sessions begin with a stimulation tolerability assessment where the dose of therapy is selected. A sham stimulation dosage will follow for the remaining procedure, including the priming stimulation, period and the standard of care rehabilitation
  Interventions: Other: Upper Limb Rehabilitation; Other: Sham Stimulation

INTERVENTIONS:
Device: NeuraStasis Stimulator System (Non-Invasive Trigeminal and Vagus Nerve Stimulation) — Pulsed electrical stimulation of the trigeminal and vagus nerves paired with upper limb rehabilitation movements
  Other Names: nTVNS
  Arms: Paired nTVNS Stimulation
Other: Upper Limb Rehabilitation — Rehabilitation movements to improve upper limb function after stroke
Other: Sham Stimulation — Control sham stimulation of the trigeminal and vagus nerves is delivered at the start of each session. Performed alongside standard-of-care rehabilitation.
  Arms: Sham Stimulation

SUMMARY:
This is a single-center, pilot study of up to 25 subjects with residual upper extremity deficits at least six months after an ischemic stroke. The purpose of the study is to evaluate the initial clinical safety, device functionality, and treatment effect of non-invasive electrical stimulation of the trigeminal and/or vagus nerves (nTVNS) using the NeuraStasis Stimulator System adjunctive to rehabilitation. Subjects will either receive the intervention or control-sham stimulation. The study will inform the design and implementation of a pivotal study.

DETAILED DESCRIPTION:
This pilot study will proceed in two phases: Phase I, an unblinded blinded stage and Phase II, a blinded stage comparing intervention and sham groups.

Phase I will consist of 5 subjects, unblinded, receiving nTVNS. This phase will test the usability of the device and de-risk the use of nTVNS during rehabilitation. Visits will include consent and baseline evaluation followed by 6 weeks of treatment consisting of the standard of care with nTVNS. Rehabilitation and treatment will occur at a cadence of 3 sessions per week. Primary endpoints will be collected after 6 weeks.

Phase II will consist of a Prospective Randomized Open, Blinded Endpoint (PROBE) design. Subjects will be randomized to an intervention nTVNS group or a control sham stimulation group. The control sham stimulation consists of standard-of-care rehabilitation with only a minimal amount of nTVNS delivered at the start of each session during a tolerability assessment intended to support further blinding for therapists and subjects. The same evaluations, sessions, and endpoints will occur as those in Phase I.

ELIGIBILITY:
Inclusion Criteria:

* History of unilateral supratentorial ischemic stroke that occurred at least 6 months but not more than 10 years prior to enrollment.
* Age >40 years and <80 years.
* Fugl-Meyer Assessment, Upper Limb (FMA-UE) baseline score of 20 to 50 (inclusive of 20 and 50).
* Ability to communicate, understand, and provide appropriate consent. Subjects should be able to follow two-step commands.
* Right- or left-sided weakness of the upper extremity.

Exclusion Criteria

* Participant has implanted metallic or electronic devices in the head or neck
* Hemorrhagic stroke or a heterogenous lesion etiology
* Participant has a cardiac pacemaker or implanted or wearable defibrillator
* Participant skin in the stimulation area has open wounds, skin eruptions, swollen, infected, or inflamed areas, or skin abnormalities that could be cancerous
* Advanced cardiac, pulmonary, liver, kidney dysfunction or blood system disease
* Participant has a fever or shows clinical signs concerning for an infectious disease
* Other neurologic or musculoskeletal diseases that could interfere with the assessments of this study
* Low heart rate (<60 bpm) from a cardiac conduction block or related etiology
* Participant has a history of trigeminal neuralgia
* Participant has a history of Bell's Palsy
* History of cranial nerve neuropathy (including facial nerve injury), carotid surgery, vagotomy, or other surgical intervention on the vagus nerve
* History of recurrent syncopal events
* Known or newly-discovered aneurysm or arteriovenous malformation
* Patients who have any terminal illness such that the patient would not be expected to survive more than 90 days
* Botox injections 12 weeks prior to or during therapy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment, Upper Limb (FMA-UE) Average Change | Within 7 days of completing 6 weeks of rehabilitation
  The Fugl-Meyer Assessment, Upper Limb (FMA-UE) will be analyzed for the difference in average change after 6 weeks of therapy compared to baseline. The FMA-UE is a common scale used to measure motor impairment after a stroke. The range is 0 (more impairment) to 66 (no impairment).

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) Average Change | Within 7 days of completing 6 weeks of rehabilitation
  The ARAT will be analyzed for the difference in average change after 6 weeks of therapy compared to baseline. The ARAT is a widely used clinical scoring tool for stroke rehabilitation. The test consists of 19 items that are grouped into four sub-tests: grasp, grip, pinch, and gross movement. The total score on the ARAT ranges from 0 to 57, with a higher score indicating better performance.
Fugl-Meyer Assessment, Upper Limb (FMA-UE) Response % | Within 7 days of completing 6 weeks of rehabilitation
  The FMA-UE will be analyzed for the % of subjects that responded to treatment defined as achieving an effect equivalent to a greater than the minimal clinically important difference.
Proportion of subjects completing all pre-specified treatment doses | Upon completion of 6 weeks of rehabilitation
  Proportion of subjects completing all pre-specified treatment sessions across the 6 weeks of rehabilitation
Subject Questionnaire on Device Usage | Upon completion of 6 weeks of rehabilitation
  A questionnaire that evaluates subjects' level of comfort during use of the device on a 5-point scale, with 5 being the most comfortable and 1 being the least comfortable.
Therapist Questionnaire on Device Usage | Upon completion of 6 weeks of rehabilitation
  A questionnaire that evaluates the ease of use of the device by therapists during the administration of rehab with the device on a 5-point scale, with 5 being the most usable and 1 being the least usable.
Serious adverse device effects (SADE) rate at 24 hours post-therapy session | Up to 24 hours after each therapy session and ending 24 hours post-last therapy session at 6 weeks of rehabilitation
  SADE rate at 24 hours post-therapy sessions
Stroke impact scale (SIS) Summative Score Average Change | Within 7 days of completing 6 weeks of rehabilitation
  The Stroke Impact Scale (SIS) is a multidimensional self-reported measure of health-related quality of life. The SIS includes 59 items and assesses 8 domains: strength (four items), memory and thinking (seven items), emotion (nine items), communication (seven items), activities of daily living (ten items), mobility (nine items), hand function (five items) and participation and function in life activities (ten items). Each item is rated using a 5-point Likert-type scale (1 = an inability to complete the item; 5 = no difficulty experienced at all) and a global score is calculated as a summative score of each domain, transformed into a 0-100 scale. It includes an extra question on the person´s perceived stroke recovery measured in the form of a visual analogue scale from 0-100. The summative score will be analyzed for the difference in average change after 6 weeks of therapy compared to baseline.
Analysis of the number of stimulations per therapy session | Upon completion of 6 weeks of rehabilitation
  The number of paired stimulations initiated each rehabilitation session will be analyzed to understand personalized effectiveness and responder likelihood.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Savitz, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Kirt Gill, MD, Study Director — NeuraStasis, Inc
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No